CLINICAL TRIAL: NCT02027675
Title: Meal-Exercise Challenge and Physical Activity Reduction Impact on Immunity and Inflammation
Acronym: MERIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MERIIT project
Record Dates: First submitted 2013-12-19; First posted 2014-01-06 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2014-11

CONDITIONS: Asthma; Obesity
Keywords: exercise; immune function; inflammation; immunity; diet; obesity; asthma
MeSH Terms: conditions — Asthma; Obesity; Motor Activity; Inflammation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meal Exercise Challenge- Order 2 (Experimental): Two different meals,an high fat micronutrient poor meal and Mediterranean Meal will be followed by an exercise challenge and performed at different orders accordingly to the cross over design.
  Interventions: Other: High fat poor micronutrient meal; Other: Mediterranean meal
- Meal Exercise Challenge- Order 1 (Experimental): Two different meals,an high fat micronutrient poor meal and Mediterranean Meal will be followed by an exercise challenge and performed at different orders accordingly to the cross over design.
  Each arm corresponds to a different intervention order.
  Interventions: Other: High fat poor micronutrient meal; Other: Mediterranean meal

INTERVENTIONS:
Other: High fat poor micronutrient meal — The meal will be prepared by a team of nutritionist in order to comply with the demand characteristics of an high fat poor micronutrient meal.
Other: Mediterranean meal — The meal will be prepared by a team of nutritionist in order to comply with the demand characteristics of an Mediterranean meal

SUMMARY:
In a society where exercise is prescribed by physicians to increase physical condition, improve dietary habits and reduce cardiovascular risk, the impact of exercise, acute or chronic, and diet in inflammation and immunity is unknown. Specific populations can have different responses towards acute and chronic exercise. Moreover specific conditions, like the type of meal ingested, can interfere with these responses. The true effect of pre-competitive meal exercise in the immunity and inflammatory response is unknown. Acute physical inactivity periods, commonly happens during daily life, related to work or acute illness. New evidence points out that it induces immediate metabolic and endocrinological changes, these can might also be associated with changes in immune response.

Aims of this project are:

1. to assess the effect of the precompetitive meal on the inflammatory, neuro-immune and metabolic response to exercise;
2. to assess the effects of sedentary behaviour on inflammatory, neuro-immune and metabolic response;
3. to assess differences in changes between healthy, asthmatic and obese subjects

DETAILED DESCRIPTION:
Two interventions will be performed for assessing the research questions and aims:

A) Randomized cross-over, with a wash out period of 7 days, single-blinded trial where two different pre-competitive meals will be followed by an exercise challenge; inflammatory neuro-immune and metabolic response will be assessed before and after each challenge.

Participants will be recruited from advertisement and four different groups will be compared: obese-asthmatic; asthmatic non-obese; obese without asthma and non-asthmatic and non-obese. All patients will be allocated to a meal challenge in which a high fat poor micronutrient meal followed by a Mediterranean meal or vice-versa; meal challenge order will be randomized and participants will be blinded to the intervention. The main outcome for this intervention will be airway inflammation and lung function. All outcomes will be assessed before and 3h after each meal.

A group of individuals will, in the three hours after the meal, perform an exercise challenge, which is aimed to induce acute immune changes.

B) Randomized controlled trial where participants, after a run-in period and eligibility evaluation, will be allocated to an intervention consisting in a reduction of physical activity by 50% or maintaining habitual physical activity for two weeks; inflammatory neuro-immune and metabolic response will be assessed before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* controlled mild to moderate asthma;
* Body mass index (BMI) ≥ 25 kg/m2; healthy participants (non asthmatic with a BMI 18,5 to 25 kg/m2) will be used for comparison;

Exclusion Criteria:

* respiratory disease other than asthma;
* severe asthma according to Global Initiative for Asthma (GINA) guidelines
* occurrence in previous 4 weeks of screening of upper/lower respiratory tract infection;
* smoking in the past 6 months and requiring mechanical ventilation for respiratory event within 6 months of screening.
* Medical conditions (hematologic, cardiovascular, renal, hepatic, neurologic or metabolic) or medication that may interfere with meal or physical activity intervention;
* Significant chronic infectious diseases (eg, HIV, hepatitis B or C);
* Abnormal electrocardiogram screening, cardiac arrhythmia, angina, congestive heart failure; renal or hepatic failure and systemic disease, mal-absorption disease history or intestinal inflammatory disease;
* Women breast-feeding, pregnant or intending pregnancy during study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Airway inflammation | Up to 6 months
  1. Lung function before and after challenge and bronchodilator response;
  2. Exhaled nitric oxide;
  3. Exhaled breath condensate (EBC);

SECONDARY OUTCOMES:
Autonomic nervous system response | Up to 6 months
  Rest heart rate; pupillary response, before and after challenge Neuropeptides measurement
Oxidative stress biomarkers | Up to 6 months
  Assessment of plasma F2-isoprostanes, lipid hydroperoxides, protein carbonyls, hydrogen peroxide and lipid soluble antioxidants
Circulating blood leukocyte-total and differential leukocyte counts and lymphocyte subpopulations assessment. | Up to 6 months
  Evaluated by flow cytometry: T cell (CD4+/CD8+), and their subsets; B cells (CD19+), Natural Killer (NK) cells (CD16+/56+), their subsets; monocytes subsets; oxidative burst activity

OTHER OUTCOMES:
Histamine skin test reactivity | Up to 6 months
  Histamine skin test reactivity, assessed by skin prick test response

CONTACTS AND LOCATIONS:
Overall Officials: Diana Silva, MD, Principal Investigator — Faculty of Medicine of Porto University; Rita Moreira, Principal Investigator — Faculty of Nutrition and Food Sciences of the University of Porto
Locations (3):
- Portugal (3):
  - Faculty of Nutrition and Food Sciences of the University of Porto, Porto, Porto District
  - Faculty of Sports of Porto University, Porto, Porto District
  - Faculty of Medicine of Porto University, Portugal, Porto District

REFERENCES:
- See also: Related Info — http://meriitproject.weebly.com/